CLINICAL TRIAL: NCT06624644
Title: A Multicenter, Open-Label, Randomized, Controlled Study to Assess the Antitumor Activity of LNS8801 With and Without Pembrolizumab in Patients With Treatment-Refractory, Unresectable Melanoma
Brief Title: A Trial of LNS8801 With or Without Pembrolizumab in Patients With Refractory Melanoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Linnaeus Therapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNS-103
Record Dates: First submitted 2024-09-27; First posted 2024-10-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Melanoma (Skin Cancer); Melanoma Stage IIIB-IV; Cutaneous Melanoma; Unresectable Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Drug Therapy; Dacarbazine; Temozolomide; Immunotherapy; Nivolumab; relatlimab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1:1 between LNS8801 + pembrolizumab, LNS8801 monotherapy, and PC arms. In the LNS8801 + pembrolizumab arm, LNS8801 will be administered every day per week and pembrolizumab will be administered 200 mg Q3W for up to 35 cycles (approximately 2 years; Note: Physicians may modify the pembrolizumab regimen to 400 mg Q6W pembrolizumab after 6 months of treatment, if appropriate). In the monotherapy arm, LNS8801 will be administered every day per week. In the PC arm, patients may receive chemotherapy (dacarbazine, temozolomide) or immunotherapy (pembrolizumab, nivolumab/relatlimab, nivolumab/ipilimumab). Patients' randomization will be stratified by normal or elevated baseline LDH, number of disease sites (<3 or ≧3), and physician's determination of primary vs secondary resistance to prior anti-PD-1 therapy per SITC guidance. Patients who are on LNS8801 + pembrolizumab combination therapy may drop one of the study medications for safety reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- LNS8801 Monotherapy (Experimental): 125 mg LNS8801 by mouth every day
  Interventions: Biological: LNS8801
- LNS8801 + Pembrolizumab (Experimental): 125 mg LNS8801 by mouth every day plus 200 mg Pembrolizumab by IV infusion once every 3 weeks.
  Interventions: Biological: LNS8801; Biological: Pembrolizumab
- Physician's Choice (Active Comparator): patients may receive chemotherapy or immunotherapy as determined by physician.
  Interventions: Drug: Chemotherapy (dacarbazine or temozolomide); Biological: Immunotherapy (Pembrolizumab); Biological: Immunotherapy (nivolumab and relatlimab); Biological: Immunotherapy (ipilimumab and nivolumab)

INTERVENTIONS:
Biological: LNS8801 — G protein-coupled estrogen receptor (GPER) agonist
  Arms: LNS8801 + Pembrolizumab; LNS8801 Monotherapy
Biological: Pembrolizumab — Recombinant monoclonal antibody (anti-PD1)
  Arms: LNS8801 + Pembrolizumab
Drug: Chemotherapy (dacarbazine or temozolomide) — chemotherapy (dacarbazine, temozolomide)
  Arms: Physician's Choice
Biological: Immunotherapy (Pembrolizumab) — pembrolizumab
  Arms: Physician's Choice
Biological: Immunotherapy (nivolumab and relatlimab) — nivolumab and relatlimab
  Arms: Physician's Choice
Biological: Immunotherapy (ipilimumab and nivolumab) — ipilimumab and nivolumab
  Arms: Physician's Choice

SUMMARY:
The goal of this clinical trial is to understand if a new drug called LNS8801 can safely treat patients with melanoma. The primary question to be answered is what is the average length of time during which melanoma does not grow or spread after starting treatment with LNS8801? Researchers will compare LNS8801 taken alone or LNS8801 taken together with another drug called pembrolizumab to other therapies as decided by the treating doctor.

135 patients will be randomly (like flipping a coin) placed in 3 treatment groups.

In the first group (LNS8801 only) - Patients will take 125mg tablet of LNS8801 by mouth once per day every day for up to 2 years.

In the second group (LNS8801 + pembrolizumab) - Patients will take 125mg tablet of LNS8801 by mouth once per day plus 200 mg of pembrolizumab by IV infusion once every 3 weeks for up to 2 years.

In the third group, called Physician's Choice (PC), patients will receive chemotherapy (dacarbazine or temozolomide) or immunotherapy (pembrolizumab, nivolumab/relatlimab or nivolumab/ipilimumab) as determined by their treating physician.

How often the patient visits the clinic visits will depend on the treatment group. Besides returning to the clinic for treatment, the patient will undergo periodic safety assessments and other required study procedures such as imaging assessments.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, multicenter study to characterize the safety, tolerability, and antitumor effects of LNS8801 alone and in combination with pembrolizumab in treatment refractory, unresectable cutaneous melanoma patients who are homozygous for the consensus GPER protein-coding amino acid sequence (C/C) and have progressed on prior immune checkpoint inhibitor therapy, including an anti-PD-1 therapy. The C/C form of GPER is present in approximately 55% of patients.

Patients must initially consent to a prescreening blood-based genetic test only. Patients with the required genotype will then consent to full screening and treatment, and the potential physician's choice (PC) treatment will be identified. Patients will be randomized 1:1:1 between LNS8801 + pembrolizumab, LNS8801 monotherapy, and PC treatment. In the LNS8801 + pembrolizumab arm, LNS8801 will be administered every day per week, and pembrolizumab will be administered 200 mg Q3W for up to 35 cycles (approximately 2 years; Note: Physicians may modify the pembrolizumab regimen to 400 mg Q6W pembrolizumab after 6 months of treatment if appropriate). In the monotherapy arm, LNS8801 will be administered every day per week. In the PC arm, patients may receive chemotherapy (dacarbazine, temozolomide) or immunotherapy (pembrolizumab, nivolumab/relatlimab, nivolumab/ipilimumab).

Patients' randomization will be stratified by normal or elevated baseline LDH, <3 or ≥3 disease sites, and physician's determination of primary vs secondary anti-PD-1 therapy resistance per SITC guidelines; prior to randomization, the preferred PC treatment for each patient will be identified, and the patient must be willing to receive this therapy if assigned to the PC arm. At least one-third of patients in each arm must have had secondary resistance to prior anti-PD-1 therapy. Patients who are on LNS8801 + pembrolizumab combination therapy may drop one of the study medications and continue on the other for tolerability or safety reasons. For example, if a patient has an immune-related AE that warrants discontinuation of pembrolizumab, they should continue LNS8801 monotherapy. Patients may choose to remain on study drugs past progression if they are clinically stable and the treating physician believes that continued therapy is likely to benefit the patient.

Patients may continue on LNS8801 therapy past progression and initiate localized therapy if they are clinically stable and the treating physician believes that continued LNS8801 therapy is likely to benefit the patient. Safety assessments will be performed on all patients at screening, throughout their participation in the study, and at either 30 days following the last dose of study drugs if they are not taking an immune checkpoint inhibitor (ICI) or 90 days following the last dose if their treatment included an ICI. Measures of metabolic health (eg, circulating lipids, blood pressure, HbA1C) will also be recorded throughout the study.

Overall survival and reason for mortality should be assessed after the last dose of study medication, every 6 months for the first year, and then annually, until it has been 2 years since any patient has taken study medication. Any anti-cancer therapies should be recorded.

Imaging of tumors for evidence of tumor response and/or progression will be performed at screening (within 21 days of the first dose of study drug) and then every 8 weeks for the first year, every 12 weeks for the second year, and every 6 months thereafter.

Up to 135 patients will be randomized in this study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed unresectable and/or metastatic cutaneous melanoma.
* 2 copies of the fully functional form of GPER protein-coding sequence.
* Eligible for and willing to receive 1 or more of the physician's choice (PC) therapies.
* Able to swallow tablets.
* Progressed on treatment with an anti-PD-1 monoclonal antibody (mAb) administered either as monotherapy or in combination with other therapies.
* Received an anti-CTLA-4 and/or BRAF containing regimen or is not eligible for or has declined anti-CTLA-4 and/or BRAF therapy prior to and for this study.
* Measurable disease.
* Eastern Cooperative Oncology Group Performance Status of 0 to 1.

Exclusion Criteria:

* Blue nevus subtype, mucosal, acral lentiginous, or uveal/ocular/choroidal Melanoma.
* Previous anti-cancer or investigational drug/device treatment within 4 weeks of the first dose of study drug.
* Radiotherapy within 2 weeks of starting study drug.
* Allogeneic tissue/solid organ transplant.
* Unstable autoimmune or immunodeficiency disease.
* Other concurrent health issues that would make participation or completion of the study difficult.
* Prior reaction to anti PD-1 therapy that would make treatment with pembrolizumab unadvisable.
* Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Compare progression-free survival (PFS) of LNS8801 + pembrolizumab vs PC arms as assessed by RECIST v1.1. | up to 2 years.
  Compare PFS between each of the 3 arms

SECONDARY OUTCOMES:
Overall Survival (OS) of LNS8801 + pembrolizumab with PC treatment | up to 5 years after the end of treatment
  Median OS compared between each of the 3 arms.
Hospitalization days of LNS8801 + pembrolizumab vs LNS8801 monotherapy vs PC arms. | Length of hospital stay (assessed up to 10 days)
  compare length of hospital stays between each of 3 arms
Duration of Response (DOR) of LNS8801 + pembrolizumab vs LNS8801 monotherapy vs PC arms. | up to 2 years.
  Duration partial response or complete response by RECIST v1.1. DOR compared between each of the 3 arms
Overall Response Rate (ORR) of LNS8801 + pembrolizumab vs LNS8801 monotherapy vs PC arms. | up to 2 years
  ORR is defined as partial response or complete response by RECIST v1.1. ORR compared between each of the 3 arms
Duration of Disease Control (DDC) of LNS8801 + pembrolizumab vs LNS8801 monotherapy vs PC arms. | up to 2 years.
  Duration of stable disease, partial response, or complete response by RECIST v1.1. DDC compared between each of the 3 arms
Percent of patients experiencing treatment-emergent adverse events and serious adverse events in LNS8801 + pembrolizumab vs LNS8801 monotherapy vs PC arms. | Duration of Treatment (up to 2 years)
  TEAE and SAE compared between each of the 3 arms
PFS of LNS8801 monotherapy vs physician's choice treatment using RECIST 1.1 | up to 2 years.
  PFS compared between 2 arms
PFS of LNS8801 monotherapy vs LNS8801 + pembrolizumab using RECIST 1.1 | up to 2 years.
  PFS compared between arms
Disease Control Rate (DCR) of LNS8801 + pembrolizumab vs LNS8801 monotherapy vs PC arms. | up to 2 years.
  Time to stable disease, partial response, or complete response by RECIST v1.1 DCR compared between each of the 3 arms

OTHER OUTCOMES:
OS in patients treated beyond progression vs those who stopped treatment at progression. | up to 5 years after the end of treatment
  Median OS compared between patients treated beyond progression and those who stopped treatment without progression.
Change in quality of life (QOL) survey responses during therapy (QLQ-C30 questionnaire) on therapeutic intervention in LNS8801 + pembrolizumab vs LNS8801 monotherapy vs PC arms. | At the beginning of Cycle 1 (each cycle 6 weeks), 2, and 3 then every 12 weeks for 1 year
  Compare between each of the 3 arms
Subgroup analyses comparing patients with primary vs secondary resistance to prior PD-1 therapy, LDH, and extent of disease. | Collected at screening
  Patients will be stratified by normal or elevated baseline LDH, less than 3 or ≧3 disease sites, and physician's determination of primary vs secondary anti-PD-1 therapy resistance as per SITC guidance
Changes in overall health measures (blood pressure). | Screening visit 2 and every 6 weeks up to on average 2 years.
  Blood draw collected at screening and then every 6 weeks starting with Cycle 1.
Changes in overall health measures (circulating lipids). | Screening visit 2 and every 6 weeks up to on average 2 years.
  Blood draw collected at screening and then every 6 weeks starting with Cycle 1.
Changes in overall health measures ( HbA1C). | Screening visit 2 and every 6 weeks up to on average 2 years.
  Blood draw collected at screening and then every 6 weeks starting with Cycle 1.
Time to new treatment or death (TNTD) of LNS8801 + pembrolizumab combination therapy vs LNS8801 monotherapy vs PC arms. | up to 2 years
  TNTD compared between each of the 3 arms
PFS in patients who received therapy for at least 2 weeks without dose holidays greater than 14 days between evaluations. | up to 2 years.
  Evaluation of PFS in patients who did not experience a dose holiday greater than 14 days
Percent of patients experiencing treatment-emergent adverse events (TEAE) and serious adverse events potentially related to therapeutic intervention in LNS8801 + pembrolizumab vs LNS8801 monotherapy vs PC arms. | up to 51 months
  Patients experiencing adverse events will be documented up to 90 days after the end of study treatment.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - USC Newport Beach, Newport Beach, California
  - UCSF, San Francisco, California
  - Stanford, Stanford, California
  - University of Colorado Anschutz, Aurora, Colorado
  - Dana Farber, Boston, Massachusetts
  - University of New Mexico, Albuquerque, New Mexico
  - UPenn, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No